CLINICAL TRIAL: NCT04508283
Title: Fiber Intake Profile Among Children 6-36 Months in Relation to Type of Milk Consumption, Gastrointestinal Symptoms and Iron Status: a Cross-sectional Study in Jakarta and Bandung, Indonesia
Brief Title: Fiber Intake Among Children in Relation to Milk Type, Gastrointestinal Symptoms and Iron Status: a Cross-sectional Study
Status: Completed | Type: Observational
Sponsor: Indonesian Nutrition Association (Other)
Responsible Party: Sponsor
Other Study IDs: INA/FI-20040450
Record Dates: First submitted 2020-08-04; First posted 2020-08-11 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Healthy Children

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fiber as part of the plants can be provided through eating grains, fruits and vegetables. As source of fiber, exclusively breastfed infants do not need additional dietary fiber because breast-milk provides oligosaccharides to maintain the bulk for normal gastrointestinal movements together with gut probiotics. However, after the period of six months of exclusive breastfeeding, then complementary foods are the initial sources of fiber of children aged 6-59 months diet, e.g. cereals, fruits and legumes should then be introduced. However, investigators should consider on the effect of plant foods as a non-haem iron food source that is less bioavailable for iron absorption. There are other dietary factors that inhibit iron bioavailability, i.e. phytates in grains and rice, vegetables protein, calcium and phosphorus in cow's milk and cheese. iron deficiency is remained common globally, especially for children age 6-24 month in which it can developing into a severe condition, i.e. iron deficiency anemia. Iron deficiency as well as anemia is closely related to delay child growth and development, negatively associated with height-for-age, and anemia are at risk for poorer cognitive, motor, social-emotional, and neurophysiologic development in the short- and long-term outcome. The aim of this study is to see the association between fiber intake from different type of milk consumption sources and dietary habits to gastrointestinal health, anemia and growth status among children aged 6-36 months.

DETAILED DESCRIPTION:
This study is an observational cross-sectional study to get fiber intake profile among children aged 6-36 months in relation to cow's and non-cow's milk consumption, gastrointestinal symptoms, hemoglobin value and nutritional status. The participants in this study are children aged 6-36 months who are recruited from selected Puskesmas (Health Care Center) in Jakarta and Bandung after provided with informed consent from children's parents. To get proportion of low fiber intake with a degree of reliability 95% and significance level of 5%, then 400 subjects is needed as a minimal sample size in this study.

The children's parents will be interviewed about socio-demographic characteristics of the subjects, gastrointestinal symptoms during the past two weeks using VAS (Visual Analogue Scale) on frequency of bowel movements in a week, parents's education, family income, and child's food intake. The children's weight and height will be measured and blood sample will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-36 months who are recruited from selected Puskesmas (Health Care Center) in Jakarta and Bandung after provided with informed consent from their parents

Exclusion Criteria:

* Children who are seriously ill and/or need special medication

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 6-36 months are recruited from selected Puskesmas (Health Care Center) in Jakarta and Bandung
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Fibre intake profile | 1 day
  Interview the parents about child's food intake using 24-hour food recall and semi-quantitative food frequency questionnaire
Type of milk consumption | 1 day
  Interview the parents about child's milk consumption
Gastrointestinal symptoms | 1day
  Interview the parents about child's gastrointestinal symptoms during the past two weeks using VAS on frequency of bowel movements in a week, the presence of difficulty when passing a bowel movement, bloating, abdominal pain/colic, and flatulence, into four scale, i.e. 0 = never, 1 = rarely, 2 = frequently, or 3 = all the time
Iron status | 1 day
  Child's blood will be taken for hemoglobin assessment
Nutritional status | 1 day
  Nutritional status will be determined using weight-for-age, height-for-age and weight-for-height indicator

CONTACTS AND LOCATIONS:
Overall Officials: Saptawati Bardosono, Doctor, Principal Investigator — Indonesian Nutrition Association
Locations (1):
- Puskesmas Kecamatan Kampung Melayu, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hermina and Prihartini. Fruits and vegetables consumption of Indonesian population in the context of balanced nutrition: A Further Analysis of Individual Food Consumption Survey (SKMl). Buletin Penelitian Kesehatan (Health Research Bulletin);2016;44(3): 205-218.
- [Background] Rakotonirainy NH, Razafindratovo V, Remonja CR, Rasoloarijaona R, Piola P, Raharintsoa C, Randremanana RV. Dietary diversity of 6- to 59-month-old children in rural areas of Moramanga and Morondava districts, Madagascar. PLoS One. 2018 Jul 13;13(7):e0200235. doi: 10.1371/journal.pone.0200235. eCollection 2018. PMID 30005067
- [Background] UNICEF. The state of the world's children: Children, food and nutrition: growing well in a changing world 2019.
- [Background] Wellington MoH. Food and Nutrition Guidelines for Healthy Infants and Toddlers (Aged 0- 2): A background paper (4th Ed) - Partially Revised December 2012
- [Background] Khan JR, Awan N, Misu F. Determinants of anemia among 6-59 months aged children in Bangladesh: evidence from nationally representative data. BMC Pediatr. 2016 Jan 11;16:3. doi: 10.1186/s12887-015-0536-z. PMID 26754288
- [Background] Widjaja IR, Widjaja FF, Sanotos LA, Wonggokusuma, Oktaviati. Anemia among children and adolescents in a rural area. Paediatr Indones 2014;54(2)
- [Background] Ntenda PAM, Chuang KY, Tiruneh FN, Chuang YC. Multilevel Analysis of the Effects of Individual- and Community-Level Factors on Childhood Anemia, Severe Anemia, and Hemoglobin Concentration in Malawi. J Trop Pediatr. 2018 Aug 1;64(4):267-278. doi: 10.1093/tropej/fmx059. PMID 28977637
- [Background] Lozoff B. Iron deficiency and child development. Food Nutr Bull. 2007 Dec;28(4 Suppl):S560-71. doi: 10.1177/15648265070284S409. PMID 18297894